CLINICAL TRIAL: NCT04905420
Title: Impact of the Pulmonary and Critical Care Medical(PCCM) Standardized Management on Healthcare Management Among Asthma or COPD or Asthma-COPD Overlap Patients: a Retrospective Descriptive Analysis (PCCM-IMPACTS)
Brief Title: The Impact of PCCM on Healthcare Among Asthma or Chronic Obstructive Pulmonary Disease (COPD) or Asthma-COPD Overlap Patients
Acronym: PCCM-IMPACTS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589BR00066
Record Dates: First submitted 2021-04-30; First posted 2021-05-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Asthma; COPD; Asthma-COPD Overlap
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Multi-centre, retrospective study describing the impact of PCCM standardized implementation on healthcare management among Asthma or COPD or Asthma-COPD overlap patients in Tianjin city of China, using real world electronic medical record database collected in local health care settings.

DETAILED DESCRIPTION:
This is a multi-center retrospective study to describe the impact of PCCM on healthcare management of Asthma or COPD or ACO patients in Tianjin healthcare big data platform database in China from Jan 01, 2015 to Dec 31, 2020. The impact of PCCM on healthcare management among Asthma or COPD or ACO patients will be explored. Analyses will be performed separately by disease, by hospitals with or without PCCM implementation, by period (pre-PCCM vs post-PCCM period) and by hospital grade. Patients enrolled into pre-PCCM period who also had post-PCCM visit(s) will be counted separately in two periods. The statistical analyses of this study will be primarily descriptive in nature and does not attempt to test any specific a priori hypotheses unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

Of note, the following criteria will be applied separately to the pre-PCCM period and post-PCCM period.

* Asthma:

  * Patients were age 18 years and older.
  * Patients had Asthma diagnosis record according to the International Classification of Disease 10th edition (ICD-10) codes J45,J45.x, J46, J46.x.
* COPD:

  * Patients were age 18 years and older.
  * Patients had COPD diagnosis record according to the International Classification of Disease 10th edition (ICD-10) codesJ44 and J44.x (including the other clinical diagnostic records for COPD diagnosis codes: the other clinical diagnostic records will be defined as chronic bronchitis or emphysema or chronic wheeze bronchitis+ at least one of the following prescribed medicine which will be defined as ICS, LABA, LAMA, ICS/LABA, LABA/LAMA, ICS/LABA/LAMA, theophylline (sustained) , systemic glucocorticoids (IV/Oral), SAMA, SABA, SABA/SAMA).
* ACO:

  * Patients were age 18 years and older.
  * Patients had both COPD and Asthma diagnosis in a single record or within one year according to the International Classification of Disease 10th edition (ICD-10) codes J44, J44.x, J45,J45.x, J46 and J46.x.

Exclusion Criteria:

* Asthma

  * Patients with any history of diagnosis of COPD.
  * Patients had new diagnosis of COPD during Asthma follow up period.
* COPD

  * Patients with any history of diagnosis of Asthma or bronchiectasis, interstitial lung disease(i.e. pulmonary fibrosis).
  * Patients had new diagnosis of Asthma during COPD follow up period.
* ACO • Patients with any history of diagnosis of bronchiectasis, interstitial lung disease (i.e. pulmonary fibrosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in analyses will be patients with at least one diagnosis of Asthma or COPD or ACO identified from the Tianjin healthcare big data platform database from Jan 01, 2015 to Dec 31, 2020. Based on the preliminary assessment, there will be around 90,000 COPD patients, 150,000 Asthma patients and 50,000 ACO patients from 8 tertiary hospitals during Jan 01, 2015 to Dec 31, 2020. In addition, approximately 1,128,890 patients attending hospital respiratory departments for all-causes from Jan 01, 2015 to Dec 31,2020.
Sampling Method: Probability Sample
Enrollment: 288538 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of newly diagnosed | Within one year
  Incidence rate of newly diagnosed (annualized) = number of newly diagnosed with disease (Asthma or COPD or ACO) /total person-time(in person-years) of patients with all-cause unique visits in respiratory department free of new Asthma or COPD or ACO diagnosis
Absolute number of Asthma or COPD or ACO patients(per ICD-10) annually | Within one year
  Absolute number of diagnosis will be defined as the number of patients with Asthma or COPD or ACO (on/after index date 1)
Proportion of Asthma or COPD or ACO patients(per ICD-10) annually | Within one year
  Prevalence of Asthma or COPD or ACO patients =total numbers with disease(Asthma or COPD or ACO) patients (on/after index date 1)/ total numbers of patients with at least one all-cause visit in respiratory department×100%
Diagnostic accordance rate of admission and discharge | Within one year
  Diagnostic accordance rate of admission and discharge = total records of accordance of admission and discharge with disease(Asthma or COPD) (on/after index date 1)/ total records of disease(Asthma or COPD) diagnosed in admission or discharge(on/after index date 1)× 100%
Proportion of prescription of inhaled medicine | Within one year
  Proportion of prescription of inhaled medicine for outpatient visits and discharges respectively
Proportion of lung function tested | Within one year
  Proportion of lung function tested= number of Asthma or COPD or ACO patients with lung function tested(on/after index date 1) /number of Asthma or COPD or ACO diagnosed(on/after index date 1) ×100%

SECONDARY OUTCOMES:
To describe demographics at baseline | Within one year
  To describe demographics among disease(Asthma or COPD or ACO) patients and disease(Asthma or COPD or ACO) patients with exacerbations history
To describe clinical characteristics at baseline | Within one year
  To describe clinical characteristics among disease(Asthma or COPD or ACO) patients and disease(Asthma or COPD or ACO) patients with exacerbations history at baseline
To describe treatment pattern at baseline | Within one year
  To describe treatment pattern among disease(Asthma or COPD or ACO) patients and disease(Asthma or COPD or ACO) patients with exacerbations history at baseline.
Proportion of standardized treatment | Within one year
  Proportion of standardized treatment=number of standardized treatment patients /number of patients with disease(Asthma or COPD or ACO) diagnosed or (disease(Asthma or COPD or ACO) patients with exacerbation history)×100%
Proportion of patients with moderate or severe Asthma or COPD or ACO exacerbation | Within one year
  Proportion of patients with moderate or severe Asthma or COPD or ACO exacerbation frequency,Asthma or COPD or ACO exacerbation frequency will be classified as follow: 0 moderate/severe,1 moderate+ 0 severe, 2 moderate+ 0 severe, ≥3 moderate+ 0 severe, 1 severe, 2 severe, ≥3 severe
Rate of exacerbations (moderate or severe) | Within one year
  Rate of exacerbations (moderate or severe) within one year after index date
Time to first moderate/severe exacerbation | Within one year
  Time to first moderate/severe exacerbation within one year after index date
All-cause mortality | within one year
  All-cause mortality within one year after the index date
Average length of stay | Within one year
  Average length of stay= total length of Asthma or COPD or ACO -related stay/total number of discharged Asthma or COPD or ACO patients.
Number of OPD, ED or inpatients visits | Within one year
  Number of OPD, ED or inpatients visits will be counted in terms of disease(Asthma or COPD or ACO)-related OPD, ED or inpatients visits
Per capita medical costs of inpatients | Within one year
  Per capita medical costs of inpatients = total medical costs(medications and non-drug treatments)/ total number of discharges.
Per capita medical costs | Within one year
  Per capita medical costs= total medical costs(medications and non-drug treatments) of Asthma or COPD-related OPD, ED or inpatients visits / total number of Asthma or CODP or ACO patients.
Average daily hospitalization medical costs | Within one year
  Average daily hospitalization medical costs=total hospitalization costs/ total length of stay of the hospitalization.
To analyze outcomes of secondary objectives separately | Within one year

OTHER OUTCOMES:
To describe demographics | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe clinical characteristics | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe treatment pattern | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe clinical outcomes | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe HRU | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe costs | Within one year
  By disease (i.e. Asthma or COPD or ACO) from Jan 01, 2014 to Dec 31, 2020.
To describe demographics | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To describe clinical characteristics | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To describe treatment pattern | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To describe clinical outcomes | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To describe HRU | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To describe costs | Within one year
  By disease (i.e. Asthma or COPD or ACO) by escalating to triple therapy or initiating triple therapy on definition of different triple therapies ) from Jan 01, 2014 to Dec 31, 2020.
To analyze outcomes of secondary objectives separately | Within one year
  To analyze outcomes of secondary objectives separately as subgroups within one year after index date

CONTACTS AND LOCATIONS:
Overall Officials: chuan Yue Li, Dr., Principal Investigator — Tianjin Chest Hospital
Locations (1):
- Tianjin Chest Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BR00066&attachmentIdentifier=3c7afbf2-3eae-46ef-a858-af66a8c8e54c&fileName=PCCM_Study_REPORT_Synopsis.pdf&versionIdentifier=